CLINICAL TRIAL: NCT00752284
Title: Randomized Controlled Trial of Safety of Coronectomy Versus Excision of Wisdom Teeth
Brief Title: Safety of Coronectomy vs Excision of Wisdom Teeth
Acronym: coronrct
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Dr Yiu Yan Leung, Oral and maxillofacial surgery, the Univeristy of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UW 06-218 T/1243
Record Dates: First submitted 2008-09-01; First posted 2008-09-15 (Estimated); Last update posted 2008-12-08 (Estimated); Status verified 2008-09

CONDITIONS: Pain; Infection; Alveolar Nerve Injury
Keywords: coronectomy; neurosensory deficit; third molar surgery
MeSH Terms: conditions — Pain; Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Coronectomy Group. Removal of crown of lower wisdom tooth, trim down root below crestal bone and primary closure
  Interventions: Procedure: Coronectomy
- B (Active Comparator): Control Group:
  total excision of lower wisdom tooth
  Interventions: Procedure: Total Excision

INTERVENTIONS:
Procedure: Coronectomy — Coronectomy Group. Removal of crown of lower wisdom tooth, trim down root below crestal bone and primary closure
  Other Names: Coronectomy Group
  Arms: A
Procedure: Total Excision — Total excision of lower third molar
  Arms: B

SUMMARY:
The purpose of this study is to compare the surgical complications and neurosensory disturbance of coronectomy and conventional excision of wisdom teeth with roots in close proximity to inferior alveolar nerve. Hypothesis: Coronectomy of wisdom tooth can reduce the chance of injury to the inferior alveolar nerve in cases of radiographic proximity to the roots when compared with conventional method of surgical removal of wisdom teeth, and there is no difference in other surgical morbidities.

DETAILED DESCRIPTION:
Complications of impacted wisdom teeth, such as pericoronitis, caries and periodontal disease are common, and these contribute to the indications that third molar surgery is still the most common oral surgical procedure performed. Damages to the inferior alveolar nerve (IAN) during surgical removal of deeply impacted wisdom teeth is a well-known complication. Over the years, reports of IAN deficit after wisdom teeth surgery were recorded from 0.4% to 8.4%. Injury to IAN can be due to compression of the nerve, either by indirect force transmitted by the root during elevation or directly by elevators. It is also possible for the nerve to be transected causing neurotmesis by rotary instruments or when the tooth is grooved or perforated by IAN. Several studies have tried to correlate radiographic markers and relationship of IAN and the root of wisdom teeth. Howe and Poyton identified 3 radiographical signs that the roots of wisdom teeth maybe grooved, notched, or perforated by the IAN 2. Rood and Shehab in 1990 suggested diversion of the canal, darkening of the root and interruption of the white line of IAN to be significantly related to IAN injury. Sedaghatfar et al. in 2005 performed a retrospective cohort study and confirmed that, and adding to it narrowing of the root to be an additional significant sign to predict the proximity of nerve and root. These radiographic signs only indicate to surgeons and patients that there is an increased risk of nerve damage associated with the removal of the corresponding wisdom tooth, but not a prevention to it if the tooth is being removed.

Coronectomy is a procedure intentionally aiming to remove only the crown of an impacted mandibular third molar, leaving the root undisturbed, and thus avoiding possible direct or indirect damage to the IAN. This technique was first described by Knutsson et al. in 1989 in a retrospective study of 33 patients. 6 more papers about coronectomy were published to date, with 3 case reports and 2 retrospective studies, and one randomized controlled trial by Renton et al. in 2005.In this last study, 128 patients were randomized to undergo either extraction or coronectomy of wisdom teeth. The group undergoing extraction was found to be significantly more common in experiencing IAN deficit after surgery than the coronectomy group, while no significant differences could be concluded in terms of other surgical morbidities. The other studies also drew similar conclusions. One common finding, however, was the slow superficial migration of the wisdom tooth root after coronectomy. It had been suggested the root is only indicated to be removed only if it is exposed intraorally, but the risk of IAN damage of the second surgery is reduced as the root has migrated away from the nerve.

ELIGIBILITY:
Inclusion Criteria:

* Radiographically the wisdom tooth root is touching or overlapping with the superior cortical line of inferior alveolar nerve or showing one or more of the following signs:

  * darkening of root
  * abrupt narrowing of root
  * interruption and loss of the white line of IAN canal
  * displacement of the IAN canal by the roots
  * Abrupt narrowing of one or both of the canal white lin

Exclusion Criteria:

* Wisdom tooth roots not touching the IAN cortical lines
* Wisdom tooth presented with apical pathology
* Pre-existing neurosensory deficit of IAN
* Systemic condition predisposing local infection: diabetes, AIDS, concurrent chemotherapy.
* Local factors predisposing infection: metabolic bone diseases e.g. fibrous dysplasia, history of radiotherapy on mandible

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 349 (Actual)
Dates: Start 2006-06; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
The incidence of neurosensory disturbance, infection or dry socket of control group and coronectomy group | 1 week-2 years

SECONDARY OUTCOMES:
Migration rate of root in coronectomy group | 1 week - 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Yiu Yan Leung, BDS, Principal Investigator — U Hong Kong; Lim Kwong Cheung, BDS, PhD, Study Director — U Hong Kong
Locations (1):
- Prince Philip Dental Hospital, Hong Kong, China